CLINICAL TRIAL: NCT01241968
Title: Randomized, Placebo Controlled, Double Blind Clinical Trial Evaluating the Treatment of Patients With Refractory Angina Pectoris With Low Intensity Extracorporeal Shockwave Therapy Device
Brief Title: Extracorporeal Shock Wave Therapy for the Treatment of Ischemic Heart Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medispec (Industry)
Collaborators: Universität Duisburg-Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESMR-RCT-DE
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Refractory Angina Pectoris
Keywords: Extracorporeal Shockwave Therapy; Myocardial Ischemia; Refractory Angina
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): A - Treatment group. Patients in this group receive actual shockwave therapy.
  Interventions: Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec)
- B (Placebo Comparator): Placebo group. This group of patients undergo the same procedure as the treatment group, however shockwaves are not delivered to the heart.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec) — Energy Density - 0.09 mJ/mm2
  Other Names: Cardiospec; ESMR therapy; Extracorporeal Shockwave Myocardial Revascularization
  Arms: A
Device: Placebo — Placebo
  Arms: B

SUMMARY:
Low intensity shockwaves have been proven in animal studies to induce local growth of new blood vessels from existing ones.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with refractory angina not amenable to revascularization with angioplasty or bypass surgery.

DETAILED DESCRIPTION:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to myocardial ischemic tissue. Shockwaves are created by a special generator and are focused using a shockwave applicator device. The treatment is guided by standard echocardiography equipment. The shockwaves are delivered in synchronization with Patient R-wave to avoid arrhythmias. The treatment is painless.

At first, the patient undergoes Stress-Echocardiography testing to identify the hypokinetic areas (ischemic areas). Following that, the ischemic areas sre treated with shockwaves. Several treatments are required for optimal results.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with chronic stable angina pectoris. Diagnosis is based on medical history, complete physical evaluation.
* Patient has documented myocardial segments with reversible ischemia.
* Patient is classified in AP CCS of III-IV.
* Patient should be on a stable dosage of medication used to treat angina for at least 6 weeks prior to enrollment.
* Patient demonstrates exercise tolerance capacity of no higher than 125 W on a modified Bruce treadmill exercise test until presence of clinical symptoms (i.e. angina, ST-depression).
* Patient demonstrates exercise tolerance time and stability averaging no more than 25% of each other (the tests will be performed within two weeks and at least a day different between the two).
* Patient has documented epicardial coronary artery disease not amenable to angioplasty or CABG.
* Patient has signed an IRB approved informed consent form.
* Patient's condition should be stable and should have a life expectancy of >12 months. Patient's current and past medical condition and status will be assessed using previous medical history, physical evaluation, and the physicians (principle investigator's) medical opinion.

Exclusion Criteria:

* Patient is pregnant
* Patient has chronic lung disease including emphysema and pulmonary fibrosis.
* Patient has active endocarditis, myocarditis or pericarditis.
* Patient is simultaneously participating in another device or drug study, or has participated in any clinical trial involving an experimental device or drug, including other drugs or devices enhancing cardiac neovascularization, or any ESWT machine of a competitor company within 3 months of entry into the study.
* Patients who are unwilling or unable to cooperate with study procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Total Exercise Time | 6 months
  The primary efficacy endpoint is the change in maximal stress exercise capacity using the modified Bruce exercise test from baseline to the 6 months post-baseline assessment.
The incidence of adverse events at 12 months post treatment | 15 months
  Incidence of patient complications, adverse reactions and rise in cardiac enzymes, blood count, platelate count renal and hepatic function, and Troponin levels, as well as E.C.G. changes, 12 months post treatment.

SECONDARY OUTCOMES:
Change in Seattle Angina Questionnaire (SAQ) | 6 months
  The change in the SAQ from baseline to 3 months post-treatment or to the last visit for patients who terminate prematurely
Change in AP-CCS | 6 months
  The AP CCS Stage at the 6 months post-baseline, or to the last visit for patients who terminate prematurely.
Change in the Number of angina attacks | 6 months
  The change in the number of angina attacks from baseline to 3 months post-treatment. The number of attacks per week will be documented.
Change in the Hospital Admission Rate | 6 months
  The change in the number of hospital admission from baseline to 3 months post-treatment. The number of attacks per week will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Lind, MD, Principal Investigator — Westdeutsches Herzzentrum ,Universität Duisburg/Essen
Locations (1):
- Westdeutsches Herzzentrum ,Universität Duisburg/Essen, Essen, Germany